CLINICAL TRIAL: NCT04623359
Title: Usefulness of High Resolution Manometry in Constipation
Acronym: MANOCOHR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2014/047/HP
Record Dates: First submitted 2020-11-04; First posted 2020-11-10 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Constipation
Keywords: high resolution manometry
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients (Experimental): Patient with constipation will have a high resolution manometry
  Interventions: Device: High resolution manometry
- Healthy volunteers (Other): Healthy volunteers will have a high resolution manometry
  Interventions: Device: High resolution manometry

INTERVENTIONS:
Device: High resolution manometry — High resolution manometry

SUMMARY:
Constipation is a frequent symptom that is reported by more than 10% of the general population. In a few case, constipation is resistant to medical standard care, including osmotic and stimulant laxatives. The diagnosis of colonic inertia may be suspected in these patients although diagnostic criteria for colonic inertia may vary from one country to another. In France, the diagnosis of colonic inertia is based on manometric study of the colorectal contractile activity using manometric probe. Using conventional manometric catheters, severe alteration of the colorectal motility is found in a very small subset of patients, who may later benefit from surgery. The recent use of high resolution manometric probe allowed to map more precisely colorectal motility, but whether these new parameters are relevant remains to be assessed. The aim of this study is to assess the diagnostic performance of a new high resolution manometric probe by comparing healthy volunteers to patients suspected of colonic inertia.

ELIGIBILITY:
For patient

Inclusion Criteria:

* Age between 18 and 65 years
* chronic Constipation (> 6 months)
* delayed colonic transit time > 100 h
* normal colonoscopy
* constipation refractory to at least 1 osmotic and 1 stimulant laxative according French guidelines on constipation ;
* Affiliated to French national healthcare insurance

Exclusion Criteria:

* Patient with constipation being either:

  * With colonic transit time <100h
  * Distal (with radio-opaque markers stasis in the rectum)
  * From organic origin
  * Recent (<6 mois)
  * Relieved using osmotic or stimulant laxatives
* Contra-indication to the use of high resolution manometry insertion

  * Intestinal occlusion
  * Coagulation disorders, including anti-coagulant treatments
  * General anesthesia contra-indication
  * colonoscopy contra-indication
* failure to perform a colonoscopy in previous attempts
* medication intake that may impair colorectal motility, including opioids
* Evolutive inflammatory of neoplasia process
* History of major digestive surgery (at exclusion of appendicectomy, cholecystectomy)
* Presence of condition that may impact digestive motility, including diabetes mellitus and sclerodermia
* Cardiologic disease that may represent a contraindication to vagal stimulation

For Healthy volunteers

Inclusion Criteria:

* Age between 18 and 65 years
* Affiliated to French national healthcare insurance

Exclusion Criteria:

* Significant digestive evolutive disease
* constipation with Kess score > 11/39 and colonic transit time ≥ 60 h
* Contra-indication to the use of high resolution manometry insertion

  * Intestinal occlusion
  * Cardiac disease
  * Coagulation disorders, including anti-coagulant treatments
  * General anesthesia contra-indication
  * colonoscopy contra-indication
* History of major digestive surgery (at exclusion of appendicectomy, cholecystectomy)
* Presence of condition that may impact digestive motility, including diabetes mellitus and sclerodermia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2023-01-25 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Frequency of isolated propagated colonic contractions | 24 hours
  Number of colonic contractions during 24 hours

SECONDARY OUTCOMES:
Speed of isolated propagated colonic contractions | 24 hours
  Average speed of colonic contractions during 24 hours
Colonic transit time | during the first 24 hours
  Transit time will be measured during during the first 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume GOURCEROL, Principal Investigator — University Hospital, Rouen
Locations (3):
- France (3):
  - CHU CAEN, Caen
  - Chu Lille, Lille
  - Rouen University Hospital, Rouen

IPD SHARING:
Plan to Share IPD: No